CLINICAL TRIAL: NCT04175613
Title: A Phase 3b, Multi Center, Open-label, Long-term Extension Study of Apremilast (CC-10004) in Pediatric Subjects From 6 Through 17 Years of Age With Moderate to Severe Plaque Psoriasis
Brief Title: A Long-term Extension Study of Apremilast (CC-10004) in Pediatric Subjects From 6 Through 17 Years of Age With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-PPSO-004; U1111-1242-3537 (Other: WHO); 2019-003497-13 (EudraCT Number)
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; CC-10004; Apremilast; Pediatric; Age 6 - 17 years
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients treated with Apremilast (Experimental): Subjects with a weight between 20 kg to < 50 kg will receive apremilast 20 mg BID and subjects with weight ≥ 50 kg at Visit 1 will receive apremilast 30 mg BID. Subjects that begin the study receiving apremilast 20 mg BID and later record a body weight ≥ 50 kg, will be switched to apremilast 30 mg BID.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast dose will be increased from 20 mg BID to 30 mg BID for those subjects that reach a weight of 50 kg or more during the study
  Other Names: CC-10004, Otezla

SUMMARY:
This study was created to provide subjects who complete Week 52 (end of Apremilast Extension Phase) of study CC-10004-PPSO-003 the option to continue to receive open-label apremilast therapy.

The study will consist of up to 208 weeks of long-term treatment followed by an 8-week observational follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

Subject must satisfy the following criteria to be enrolled in the study:

1. Subject is male or female 6 to 17 years of age, inclusive, at the time the informed consent document is signed by the legal guardian.
2. Subject must have a weight of ≥ 20 kg.
3. Subjects must have an age and sex specific BMI value no lower in range than the 5th percentile on the Centers for Disease Control (CDC) growth chart for children and adolescents.
4. Subject must have completed Week 52 (Apremilast Extension Phase) of Study CC-10004-PPSO-003.
5. Subject is able to sign an assent with a legal guardian/s who understand/s and voluntarily sign/s an informed consent prior to any study-related assessments/procedures being conducted.
6. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
7. All female subjects of childbearing potential (FCBP) must either practice abstinence from heterosexual contact or use one of the approved contraceptive options as described below while on apremilast and for at least 28 days after administration of the last dose of apremilast. For the purpose of this study, a female subject is considered of childbearing potential if she is ≥ 12 years old or has reached menarche, whichever occurred first.

At the time of study entry, and at any time during the study when a female subject of childbearing potential's contraceptive measures or ability to become pregnant changes, the Investigator will educate the subject regarding abstinence or contraception options and the correct and consistent use of effective contraceptive methods in order to successfully prevent pregnancy.

Females of childbearing potential must have a negative pregnancy test at each visit. All FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy;

OR

Option 2: Male or female condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method:

(a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

NOTE: Option 2 may not be acceptable as a contraception option in all countries per local guidelines/regulations.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has a condition, including the presence of laboratory abnormalities, or psychiatric illness, that would place the subject at unacceptable risk if he/she were to participate in the study.
2. Subject has a condition that confounds the ability to interpret data from the study.
3. Subject has evidence of skin conditions, other than psoriasis, that would interfere with clinical assessments.
4. Subject is pregnant or breastfeeding.
5. Subject has guttate, erythrodermic, or pustular psoriasis.
6. Subject has active tuberculosis (TB) or a history of incompletely treated TB.
7. Subject answers "Yes" to any question on the Columbia-Suicide Severity Rating Scale at Visit 16 of study CC-10004-PPSO-003.
8. Subject plans concurrent use of the following therapies that may have a possible effect on psoriasis.

   1. Conventional systemic therapy for psoriasis (including but not limited to cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate, thioguanine, hydroxyurea, sirolimus, sulfasalazine, azathioprine, and fumaric acid esters)
   2. Biologic therapy:

   i. Etanercept (or biosimilar) treatment ii. Adalimumab (or biosimilar) treatment iii. Other TNF or interleukin (IL)-17 blockers (such as infliximab, certolizumab pegol, secukinumab, ixekizumab, brodalumab, or their biosimilars) iv. Anti-IL-12 or anti-IL-23 treatment (such as ustekinumab, guselkumab, or tildrakizumab) c) Use of any investigational drug other than apremilast
9. Subject has prolonged sun exposure or use of tanning booths or other ultraviolet (UV) light sources.
10. Children in Care: a child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 4 years
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Collected at each study visit throughout the life of the study - up to 4 years
  Questionnaire to monitor depression, suicidal thoughts and behavior
Weight of patients treated with Apremilast | Collected at each study visit throughout the life of the study - up to 4 years
  Body weight in kg
Mean body mass index of the patient treated with Apremilast | Collected at each study visit throughout the life of the study - up to 4 years
  BMI (combined outcome of weight and height in the form of kg/m^2)
Height patients treated with Apremilast | Collected at each study visit throughout the life of the study - up to 4 years
  Height (inches or centimeters) will be collected for all pediatric subjects and descriptively summarized
Assessment of sexual maturity | Collected every 52 weeks throughout the life of the study - up to 4 years
  Sexual maturation, assessed by Tanner staging system, will be conducted for all pediatric subjects and descriptively summarized

SECONDARY OUTCOMES:
Static Physician Global Assessment (sPGA) | Collected at each study visit throughout the life of the study - up to 4 years
  is the assessment by the Investigator of the overall disease severity at the time of evaluation. The sPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an assessment of the severity of the three primary signs of the disease: erythema, scaling and plaque elevation.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (50):
- United States (13):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Johnson Dermatology Clinic, Fort Smith, Arkansas
  - First OC Dermatology, Irvine, California
  - Stanford University School of Medicine, Palo Alto, California
  - California Dermatology Institute, Thousand Oaks, California
  - Solutions Through Advanced Research Inc, Jacksonville, Florida
  - Ciocca Dermatology, Miami, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Dawes Fretzin Dermatology Group Inc, Indianapolis, Indiana
  - Wright State Physicians, Fairborn, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Driscoll Childrens Hospital, San Antonio, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Belgium (3):
  - Centre Hospitalier Universitaire Saint Pierre, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Canada (4):
  - Stollery Childrens Hospital, Edmonton, Alberta
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - Karma Clinical Trials, St. John's, Newfoundland and Labrador
  - AvantDerm, Toronto, Ontario
- Czechia (2):
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Synexus Czech sro, Prague
- France (2):
  - Cabinet du Docteur Ruer-Mulard Mireille, Martigues
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
- Soroka University Medical Center, Bear Sheva, Israel
- Italy (3):
  - Azienda Ospedaliero Universitaria Di Cagliari, Cagliari
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Padova, Padua
- Russia (14):
  - Altai State Medical University, Barnaul
  - Chelyabinsk Regional Clinical Skin and Venereal Dispensary, Chelyabinsk
  - Republican Clinical Dermatology and Venerology Dispensary, Kazan'
  - Clinical Dispensary of Dermatology and Venereology of Krasnodar Territory of the Ministry of Health, Krasnodar
  - State Scientific Center for Dermatovenereology and Cosmetology, Moscow
  - Moscow Scientific Practical Center of Dermatology Venerology and Cosmetology, Moscow
  - National Medical Research Center for Children Health, Moscow
  - LLC Medical Center Zdorovaya Semiya, Novosibirsk
  - Pierre Wolkenshtein Skin Diseases Clinic LLC, Saint Petersburg
  - Saint Petersburg State Pediatric Medical University, Saint Petersburg
  - LLC PiterKlinika, Saint Petersburg
  - Bashkiria State Medical University, Ufa
  - Yarosavl State Medical Academy, Yaroslavl
  - Ural Scientific Research Institute of Dermatovenereology and Immunopathology, Yekaterinburg
- Spain (8):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - General University Hospital of Alicante, Alicante
  - Hopsital Germans Trias I Pujol, Badalona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Marques de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com